CLINICAL TRIAL: NCT04320212
Title: Randomized Comparative Trial of Pre-surgical Lumbar Epidural Analgesia With Bilateral Erector Spinae Block for Perioperative Pain Management in Lumbar Spine Surgery
Brief Title: Lumbar Epidural Analgesia With Bilateral Erector Spinae Block for Pain Management in Lumbar Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Kamal Zahran, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: M D-82 -2019
Record Dates: First submitted 2019-12-19; First posted 2020-03-24 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Perioperative Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lumber epidural analgesia (Active Comparator): : the patient will be placed in the lateral position, Lidocaine will be given using 5 ml syringe and a 18 G Tuohy needle will be introduced in the epidural space, using the ultrasound, under strict aseptic precautions. The ultrasound probe will be placed 90 degrees into transverse orientation and slided cephalad or caudad to obtain the transverse interspinous view (TI view) 2 levels above the operation level. patient will receive 20 ml of 0.25% plain bupivacaine after negative aspiration for blood or cerebrospinal fluid. Then, the patient will be placed in prone position to start the surgical procedure
  Interventions: Procedure: lumber epidural analgesia
- erector spinae analgesia (Active Comparator): the patient will be placed in the prone position. Then, the Erector Spinae block will be given by a high-frequency linear ultrasound transducer. The Erector Spinae muscle and transverse process will be then identified, and a 18 G Tuohy needle will be advanced, using the in-plane approach, in cephalad-to-caudal direction, through the interfascial plane between the Erector Spinae and the underlying transverse process under strict aseptic precautions until the tip is deep to erector spinae muscle. The block will be performed bilaterally by injecting 40 mL of 0.25% bupivacaine (20 mL into each side)
  Interventions: Procedure: erector spinae analgesia

INTERVENTIONS:
Procedure: lumber epidural analgesia — the lumber epidural analgesia will be given after induction of general anesthesia.
  Arms: lumber epidural analgesia
Procedure: erector spinae analgesia — the erector spinae analgesia will be given after induction of general anesthesia.
  Arms: erector spinae analgesia

SUMMARY:
Surgical procedures on the spine and spinal cord are common and are performed for a wide variety of diseases. They range from minimally invasive, single-level decompression to highly complex, multi-stage extensive reconstruction. Operative procedures for degenerative spine diseases and herniated discs are most common in those under 60 years of age. While those over 60 years of age most commonly undergo spine surgery for spinal stenosis

Patients undergoing spine surgery experience severe pain in the postoperative period. Recent studies show that the incidence of acute postoperative pain following spine surgery vary from 30 to 64%. Postoperative pain may also increase morbidity and incidence of complications and prolong postoperative rehabilitation. In addition, it is a risk factor for development of chronic pain syndromes

Postoperative pain is usually treated with oral or intravenous opioids in combination with non-steroidal anti-inflammatory drugs. However, they often results in insufficient pain control and side effects such as respiratory depression, nausea, and vomiting.

Epidural anaesthesia and analgesia have been shown to be superior to intravenous analgesia. The former is better with respect to pain quality, incidence of side effects, pulmonary, cardiac, and gastrointestinal dysfunction. However, it may be associated with hemodynamic instability. Migration of the epidural catheter with unpredictable absorption of the local anaesthetics remains a challenge to the anaesthetists. The Erector Spinae block proved to be efficient in controlling post-operative pain. It is a simple interfascial plane block, published in 2016. It provides effective analgesia for 24 hours in patients undergoing lumbar spine surgery.

Therefore, a prospective, randomized study was designed to compare the analgesic and side effects of the epidural analgesia with the Erector Spinae block in patients undergoing lumbar spine surgery. To our knowledge, this is the first clinical trial that compares the Erector Spinae block with the epidural analgesia in a variety of lumbar spine surgeries.

DETAILED DESCRIPTION:
History will be taken from all patients. Age and then American Society of Anaesthesiologists' (ASA) score will be recorded.

Preoperatively patients' pain score, laboratory investigations as complete blood picture, coagulation profile, liver and renal functions will be recorded. General examination will be carried out with examination of the back to exclude infection at the injection site and anatomical deformities.

Baseline vital signs will be recorded including non-invasive measurement of systolic, mean, diastolic arterial pressures, and heart rate and oxygen saturation.

After inserting an intravenous (IV) access, the patient will be pre-medicated with midazolam in a dose 0.1 mg/kg and metoclopramide in a dose 0.1-0.2 mg/kg.

Upon arrival to the operating room, appropriate monitors (continuous pulse oximetry, electrocardiography and non-invasive blood pressure) will be placed. Then, general anaesthesia will be induced. 1.5 μg/kg fentanyl and 2 mg/kg propofol will be given. Tracheal intubation will be facilitated with 0.5 mg/kg atracurium. Anaesthesia will be maintained using isoflurane in oxygen and air. Additional doses of 0.1 mg/kg atracurium will be administrated every 30 minutes. A urinary catheter will be placed for control of diuresis. the patient will receive either lumber epidural or erector spinae analgesia according to the group randomization.

The surgical intervention will be then allowed 20 minutes after finishing the block procedure.

Failed block is defined as increase in heart rate (HR) and mean arterial blood pressure (MABP)>20% from base line with skin incision. This will be treated by 1ug /kg of fentanyl as top-up doses and increasing isoflurane concentration in case of inadequate response to fentanyl.

In case of decrease in MABP>20% from base line, the patient will receive a 500 ml ringer infusion with 5 mg ephedrine. If HR decrease to 45 beats/minute, atropine 0.5 mg will be given.

postoperative nausea and vomiting will be managed with 0.1 mg/kg ondansetron

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II patients
* Aged 18-60 years
* Undergoing elective lumbar spine decompression and fusion surgery, using the posterior approach, under general anaesthesia.

Exclusion Criteria:

* Patients with severe cardiac diseases as ischemic heart disease, rheumatic valve disorders and cardiomyopathy.
* Contraindication to neuroaxial anaesthesia e.g. patients on anticoagulants, infection at the injection site and coagulopathy
* Hypersensitivity to the local anaesthetics used.
* Patient refusal.
* Neurologic deficits in the form of sensory loss, motor weakness or preexisting pain symptoms due to neurologic diseases apart from back pain associated with the planned operation.
* Patients with previous back surgeries

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
time to first analgesic request | from the time of performance of the intervention till the first analgesic requirement during the 24 hours postoperative
  minutes

SECONDARY OUTCOMES:
The numeric rate scale (NRS) | 5 minutes after extubation,1 hour, 2 hours, 4 hours, 8 hours, 12 hours and 24 hour postoperative
  Pain will be classified as mild (NRS 0-4), moderate (NRS 5-7), and severe (NRS 8-10)
postoperative morphine consumption | 5 minutes after extubation till 24 hour postoperative
  mg
postoperative diclofenac consumption | 5 minutes after extubation till 24 hour postoperative
  mg
systolic blood pressure | every 10 minutes from skin incision to skin closure and at 2, 4 hours post operatively.
  mmHg
heart rate | every 10 minutes from skin incision to skin closure and at 2, 4 hours post operatively.
  beat per minute

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy Hospital, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided